CLINICAL TRIAL: NCT06175598
Title: Analysis of the Causes of Redo Pull-through for Recurrent Constipation and the Risk Factors Affecting the Prognosis of the Hirschsprung's Disease and Allied Disorders
Status: Completed | Type: Observational
Sponsor: Feng Jiexiong (Other)
Responsible Party: Sponsor-Investigator, Feng Jiexiong, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJ-IRB20230739
Record Dates: First submitted 2023-12-07; First posted 2023-12-19 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Surgery; Pediatric ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Acquire Aganglionosis (AA)
- Intestinal Dysmotility (ID)
- Anastomotic Complications (AC)
- Intestinal Neurodevelopmental Impairment (INI)
- Incomplete Resection of Affected Intestinal Segments (IRAIS)

SUMMARY:
The goal of this observational study is to conducted a comprehensive analysis of the factors contributing to redo- Pull-through surgery for constipation recurrence in Children who are suffering from Hirschsprun' s disease (HSCR) and its allied disorders (ADHD) . The main question[s] it aims to answer are:

1. Our study focused on the treatment and prognosis of these conditions, drawing upon 16 years of patient data and clinical experiences"
2. What are the key risk factors affecting the prognosis of recurrent constipation patients undergoing repeat PT?

ELIGIBILITY:
Inclusion Criteria:

1. Patients admitted to the department of pediatric surgery at Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, between January 2005 and December 2021;
2. HSCR and ADHD patients admitted due to "constipation recurrence" and requiring redo-PT.

Exclusion Criteria:

1. Patients undergoing staged surgeries or undergoing internal sphincterotomy;
2. Patients with concomitant severe congenital anomalies such as Down syndrome; (3) Patients with incomplete postoperative follow-up data after redo-PT.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study collected comprehensive clinical data and compiled postoperative follow-up data from patients who underwent corrective surgery for HSCR and ADHD and subsequently required redo-PT due to recurrent constipation.
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2023-12-07 (Actual); Study Completion 2023-12-07 (Actual)

PRIMARY OUTCOMES:
Participants with redo-pull-through surgery for recurrent constipation | 1990-2023
  After utilizing the terms "Hirschsprung" and "Redo pull-through" in searches across "PubMed" and "Web of Science" for references published between 1990 and 2023, and subsequent removal of duplicate and incomplete documents, we compiled clinical information from the remaining literature. This compilation facilitated a review of relevant literature on the causes of redo-PT for recurrent constipation, enabling an assessment of classification types, which we categorized into five groups: Incomplete Resection of Affected Intestinal Segments (IRAIS), Acquire Aganglionosis (AA), Intestinal Dysmotility (ID), Anastomotic Complications (AC), and Intestinal Neurodevelopmental Impairment (INI).
Participants with and without postoperative complications | through study completion, an average of 33 year
  Group the data by gender, age groups, surgical techniques, and surgical approaches. Then, calculate the number of cases with and without postoperative complications

CONTACTS AND LOCATIONS:
Overall Officials: Jiexiong Feng, PhD, Study Director — Tongji Hospital
Locations (1):
- Department of Pediatric Surgery, Wuhan, Hubei, China